CLINICAL TRIAL: NCT06130800
Title: Respiratory Sarcopenia in Institutionalized Older Adults in the Region of Murcia: Prevalence and Associated Factors
Brief Title: Respiratory Sarcopenia in Institutionalized Older Adults in the Region of Murcia
Status: Completed | Type: Observational
Sponsor: Felipe León Morillas (Other)
Responsible Party: Sponsor-Investigator, Felipe León Morillas, Investigator, Catholic University of Murcia
Organization: Catholic University of Murcia (Other)
Other Study IDs: SarcoRespi
Record Dates: First submitted 2023-10-30; First posted 2023-11-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-01

CONDITIONS: Sarcopenia; Respiratory Function Impaired
Keywords: sarcopenia; respiratory force; institutionalized elderly
MeSH Terms: conditions — Sarcopenia; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Wheelchair: The inclusion criteria to participate in the study are being in a wheelchair, preserved cognitive status and having sufficient ability to Oral occlusion for carrying out respiratory tests. The exclusion criteria are following: presence of respiratory diseases or in treatment of respiratory diseases, serious orthopedic diseases that interfere with measurements and those with a diagnosis of dementia. In addition, those who present any contraindication for carrying out the procedure will be excluded.
  of the respiratory pressure measurement tests, as established in the SEPAR guidelines. The objectives of the study and the methodology to be used will be explained to all participants.
  An information sheet will be provided and the informed consent sheet will be given to them.
- wanderers: The inclusion criteria to participate in the study are to have functional ambulation, preserved cognitive status and have sufficient ability to Oral occlusion for carrying out respiratory tests. The exclusion criteria are following: presence of respiratory diseases or in treatment of respiratory diseases, serious orthopedic diseases that interfere with measurements and those with a diagnosis of dementia. In addition, those who present any contraindication for carrying out the procedure will be excluded.
  of the respiratory pressure measurement tests, as established in the SEPAR guidelines. The objectives of the study and the methodology to be used will be explained to all participants.
  An information sheet will be provided and the informed consent sheet will be given to them.

SUMMARY:
Objectives: The objectives of this study are to describe the prevalence of respiratory sarcopenia in institutionalized older adults. Methodology: A sample of approximately 120 older adults from 5 residences located in Murcia capital will participate in the study. A prospective observational study will be carried out, with one year of follow-up, with patients who have been diagnosed with respiratory sarcopenia. Sociodemographic and clinical variables, physical function (palm grip, 5STS, 4MGS), respiratory force variables (MIP and PEF) and diaphragmatic ultrasound (thickness, shortening fraction and diaphragmatic excursion) will be measured. Descriptive statistics, univariate and multivariate logistic regression models, Cox proportional hazards model and KaplanMeier curves will be used to analyze the data from the longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* To have functional ambulation and/or wheelchair.
* preserved cognitive status.
* have sufficient ability to Oral occlusion for carrying out respiratory tests.

Exclusion Criteria:

* presence of respiratory diseases or in treatment of respiratory diseases.
* serious orthopedic diseases that interfere with measurements and those with a diagnosis of dementia.
* those who present any contraindication for carrying out the procedure will be excluded.
* of the respiratory pressure measurement tests, as established in the SEPAR guidelines.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Institutionalized elderly diagnosed with respiratory sarcopenia
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Sociodemographic | 8 MONTHS
  Sociodemographic dates
Clinical variables | 8 MONTHS
  Clinical variables will be extracted from history clinic
Palm grip strength | 8 MONTHS
  Palm grip strength will be measured with the digital hand dynamometer (Jamar©). The Participants will remain seated with the shoulder in 0° adduction; elbow flexed 90° and forearm in neutral position. Three attempts will be made and the best value will be chosen
5 SIT TO STAND | 8 MONTHS
  The 5STS test measures the time (in seconds) it takes a subject to stop 5 times from a sitting position, as quickly as possible.
4 METRES | 8 MONTS
  The gait speed test (4MGS) measures the time it takes to cross a line of 4m at normal speed.
Body composition | 8 MONTHS
  - The analysis of body composition will be carried out with the TANITA MC 780-P MA monitor, which provides information on visceral and body fat, skeletal muscle level, BMI and basal metabolism.
Respiratoy muscle force | 8 MONTHS
  To measure respiratory muscle force, the maximum respiratory pressures will be evaluated in mouth (PIM/PEM). For them we will use an inspiratory and expiratory mouth pressure monitor maximum, a module of the Datapir touch© spirometer (Sibelmed, Barcelona). The measurement will be performed by a previously trained and experienced physiotherapist, following the protocol established by the Spanish Society of Pulmonology (4-SEPAR).
Diaphragmatic ultrasound variables | 8 MONTHS
  The diaphragmatic ultrasound variables examined will be mobility, thickness and fraction of shortening. For this we will use the Esaote MyLab™ Sigma ultrasound machine (Esaote SpA, Genoa, Italy), with double probe (linear and convex).

SECONDARY OUTCOMES:
Health results | 8 MONTHS
  The health outcome variables that will be recorded over a year will be: infections respiratory diseases, visit to the emergency department, hospitalization, bedridden and/or death. This Information will be extracted from the patient's clinical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Residence of the elderly, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No